CLINICAL TRIAL: NCT01181921
Title: Phase IV Study for the Assessment of Modulating Effect of Galantamine (Reminyl PRC) on Circadian Rhythm in Patients With Moderate Alzheimer's Disease
Brief Title: The CIRCADIAN Study: Evaluation of Modulating Effect of Galantamine on Circadian Rhythm in Patients With Mild to Moderate Alzheimer's Disease
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The recruitment rate was very low (one screening failure and one early withdrawal patient)
Sponsor: Janssen-Cilag, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CR015586; GALALZ4041 (Other: Janssen-Cilag S.A., Spain); 2009-013689-18 (EudraCT Number)
Record Dates: First submitted 2010-08-12; First posted 2010-08-13 (Estimated); Results first posted 2012-08-14 (Estimated); Last update posted 2014-05-01 (Estimated); Status verified 2014-04

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer Disease; Dementia; Sleep Disorders; Galantamine; Reminyl
MeSH Terms: conditions — Alzheimer Disease; Dementia; Sleep Wake Disorders | interventions — Galantamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Galantamine (Experimental)
  Interventions: Drug: Galantamine

INTERVENTIONS:
Drug: Galantamine — Type= range, unit= mg, number= 8-24, form= capsule, route= oral use. The starting dose will be 8 mg/day for 4 weeks. Subsequently, the initial maintenance dose will be 16 mg/day for 4 weeks. Then, an increase to the maintenance dose of 24 mg/day should be considered on an individual basis after appropriate assessment.

SUMMARY:
The purpose of this study is to assess the modulating effect of galantamine on circadian rhythm in patients with moderate Alzheimer's disease.

DETAILED DESCRIPTION:
This is a pilot, single-group, interventional, prospective study including patients with moderate Alzheimer's disease, treated with galantamine. Galantamine is thought to benefit the cognitive functioning of those with Alzheimer's disease. The starting treatment dose is 8 mg/day for 4 weeks. The initial maintenance dose of galantamine is 16 mg/day. Patients should be maintained on 16 mg/day for 4 weeks. An increase to the maintenance dose of 24 mg/day should be considered on an individual basis after the appropriate assessment including evaluation of clinical benefit and tolerability. For individual patients not showing an increased response or not tolerating 24 mg/day, a dose reduction to 16 mg/day should be considered. The primary objective is the assessment of the modulating effect of galantamine (Reminyl PRC) on circadian rhythm (wake/sleep) in patients with moderate Alzheimer's disease. The secondary objective is to assess the perception of the physicians, caregivers and patients themselves on sleep-wake disorders in patients with moderate Alzheimer's disease before and after treatment with galantamine. Sleep disturbances will be assessed by two actigraphy measures: one, before starting treatment, and the other, 12 weeks after the first actigraphic measure. The primary endpoint is the day/night ratio measured by the actigraphy before and after treatment with galantamine in patients with moderate Alzheimer-type dementia. Concerning the Efficacy Measures, the Actigraphy will be used as a method to assess the modulating effect of galantamine on circadian rate. The impact of this modulating effect on the caregivers, patients themselves and physicians will be assessed by three questionnaires: the Zarit Caregiver Burden Interview (ZBI), the Pittsburgh Sleep Quality Index (PSQI) and the Clinical Global Impression (CGI), respectively. Patient safety will be monitored. It is estimated that the study period will range from September 2010 to the second quarter of 2011.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Alzheimer-type dementia according to the definition of the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM IV-TR) and a diagnosis of possible or probable Alzheimer-type dementia, according to NINCDS-ADRDA classification (American Psychiatric Association, 2000
* McKhann, G. et al, 1984)
* should have moderate dementia, evidenced by a Mini-Mental Status examination (MMSE) score between 12 and 20, including these limits
* At inclusion, a recent CT or MRI must be available
* Physical examination and the electrocardiogram (ECG) performed at the screening visit must be normal or consistent with the underlying illness in the study population
* History of sleep behavior changes (eg: insomnia, daytime sleepiness, changes in sleep/wakefulness cycle) 2 or more weeks before, reported by the caregiver
* Patients should have a caregiver sufficiently informed of their condition and, if possible, living with them
* Patients (or their legally-acceptable representatives) must have signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study

Exclusion Criteria:

* History of other neurodegenerative disorders, such as Parkinson's disease, Pick disease or Huntington's chorea, Down syndrome, Creutzfeldt-Jakob disease (patients with mild extrapyramidal signs for which no treatment is required are not excluded from the trial)
* Clinically significant cardiovascular disease expected to limit the ability of the patient to participate and complete the study
* Any history of epilepsy or seizures (except for febrile seizures in childhood)
* Clinically significant psychiatric condition, according to the DSM-IV criteria, particularly major depression or schizophrenia currently
* Active peptic ulcer (treatment of the disease started < 3 months or treatment is not successful
* Clinically significant liver, renal, pulmonary, metabolic, or endocrine disorders
* Clinically significant urinary flow obstruction
* History of or suspected alcoholism or drug abuse in accordance to the DSM-IV criteria, in the past year, or previous history of prolonged abuse
* Previous therapy with memantine or an acetylcholinesterase inhibitor (including galantamine)
* Patients receiving antipsychotics, hypnotic or sedative agents (those patients who need this kind of medication during the study would be withdrawn from the study and replaced)
* Bedridden patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2011-05; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag S.A. (formerly Janssen Sp) Clinical Trial, Study Director — Janssen-Cilag, S.A.
Locations (1):
- Barcelona, Spain

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Only one participant was recruited and did not complete the study; therefore no assessments have been conducted throughout the study.
Groups:
- Galantamine: Galantamine (capsules/oral use). Starting dose: 8 mg/day for 4 weeks; initial maintenance dose: 16 mg/day for 4 weeks; then, an increase to the maintenance dose of 24 mg/day should be considered on an individual basis after appropriate assessment.
Period: Overall Study
Arm/Group | Galantamine
Started | 1
Completed | 0
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Galantamine
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Sleep/Wake Patterns as Measured by Actigraph at 12 Weeks
Description: Actigraph is a small portable device that is worn on the wrist of the non-dominant arm to measure body movement during long time periods. It creates a pattern based on activity that is useful in assessing sleep-wake cycles across many consecutive days and nights. It is useful for assessing sleep phase disorders.
Time Frame: Baseline and 12 weeks
Population: Only one participant was recruited and did not complete the study; therefore no assessments have been conducted throughout the study.
Arm/Group | Galantamine
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Galantamine
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Study results as well as all reports or publications related to the study, belong to the sponsor exclusively. If the investigator would like to public results in journals or scientific magazines, it has to be in agreement with the sponsor and according to the protocol.